CLINICAL TRIAL: NCT00877448
Title: A Phase I/II, Randomized, Single-Blind, Placebo-Controlled Escalating Double-Dose Safety Study of an Intramuscular Influenza Vaccine (Multimeric-001) Injected to Healthy Volunteers
Brief Title: A Double-Dose Safety Study of An Influenza Vaccine (Multimeric-001)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BiondVax Pharmaceuticals ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BVX002
Record Dates: First submitted 2009-01-28; First posted 2009-04-07 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: INFLUENZA; VACCINE; UNIVERSAL; SAFETY
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Multimeric-001 250 Mcg (Experimental): Multimeric-001 250 Mcg in PBS
  Interventions: Biological: Adjuvanted Multimeric-001 250 Mcg
- Adjuvanted Multimeric-001 250 Mcg (Experimental): 250 Mcg in montanide
  Interventions: Biological: Multimeric-001 250 Mcg
- Phosphate Buffered saline (Placebo Comparator): Non-adjuvanted placebo
  Interventions: Biological: Phosphate Buffered saline
- Adjuvanted PBS (Placebo Comparator): Adjuvant was montanide
  Interventions: Biological: Adjuvanted PBS
- Multimeric-001 500 Mcg (Experimental): Multimeric-001 in PBS
  Interventions: Biological: Multimeric-001 500 Mcg
- Adjuvanted Multimeric-001 500 Mcg (Experimental): Adjuvant was montanide
  Interventions: Biological: Adjuvanted Multimeric-001 500 Mcg
- Multimeric-001 125 Mcg (Experimental): Multimeric-001 in PBS
  Interventions: Biological: Multimeric-001 125 Mcg

INTERVENTIONS:
Biological: Adjuvanted Multimeric-001 250 Mcg
  Arms: Multimeric-001 250 Mcg
Biological: Multimeric-001 250 Mcg
  Arms: Adjuvanted Multimeric-001 250 Mcg
Biological: Phosphate Buffered saline
  Arms: Phosphate Buffered saline
Biological: Adjuvanted PBS
  Arms: Adjuvanted PBS
Biological: Adjuvanted Multimeric-001 500 Mcg
  Arms: Adjuvanted Multimeric-001 500 Mcg
Biological: Multimeric-001 500 Mcg
  Arms: Multimeric-001 500 Mcg
Biological: Multimeric-001 125 Mcg
  Arms: Multimeric-001 125 Mcg

SUMMARY:
A phase I/II, randomized, single-blind, placebo-controlled escalating double-dose safety study of an intramuscular universal influenza vaccine (Multimeric-001) injected to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 18 and 55 years (inclusive) of age.
* Non-smoking (by declaration) for a period of at least 6 months.
* Subjects able to adhere to the visit schedule and protocol requirements and be available to complete the study.
* Haematology and Chemistry values within normal ranges or with no clinical significance
* Subjects who provide written informed consent to participate in the study

Exclusion Criteria:

* Known history of significant medical disorder, which in the investigator's judgment contraindicates administration of the study medications.
* Ongoing flu symptoms or influenza
* Any clinically significant abnormality upon physical examination or in the clinical laboratory test at screening visit.
* Treatment with immune immunosuppressant drugs or other immune enhancing drugs.
* Subjects who have been immunized with anti-influenza vaccine or infected by influenza virus within one year prior to the screening visit.
* Administration of any vaccine 30 days before the screening visit.
* Known history of drug or alcohol abuse.
* Known history of HIV, hepatitis C or B virus (HCV or HBV)
* Subjects with known Guillain Barré Syndrome in the past
* 2 or more hospitalization within the last year prior to screening visit
* Increased liver enzymes 2.5 times above the upper reference level
* Known hypersensitivity and/or allergy to any drugs
* Any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
* Subjects who participated in another clinical study within 30 days prior to study entry
* Subjects who are non-cooperative or unwilling to sign consent form.
* Pregnant or lactating women at entry to study and those that are unwilling to agree to continue precautions for two months after completion of the study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, MD, Principal Investigator — Sourasky Medical Center, Tel Aviv, Israel
Locations (1):
- Tasmc Crc, Tel Aviv, Israel

REFERENCES:
- [Result] Atsmon J, Kate-Ilovitz E, Shaikevich D, Singer Y, Volokhov I, Haim KY, Ben-Yedidia T. Safety and immunogenicity of multimeric-001--a novel universal influenza vaccine. J Clin Immunol. 2012 Jun;32(3):595-603. doi: 10.1007/s10875-011-9632-5. Epub 2012 Feb 9. PMID 22318394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done on a running basis after eligibility of inclusion/exclusion criteria was met and subjects were invited to clinic after screening procedures within up to 21 days before their first vaccination.
Pre-assignment Details: After meeting eligibility criteria to enter the study subjects were randomized simultaneously.
Groups:
- Multimeric-001 250 mcg in PBS: Multimeric - 001 250 mcg in Phosphate Buffered Solution (PBS) injected twice with the interval of 21 days between them.
- Adjuvanted Multimeric -001 250 mcg: Adjuvanted Multimeric -001 250 mcg injected twice with the interval of 21 days between the injections.10 participants in total.
- PBS (Placebo): 0.2 ml of Phosphate Buffered Saline is injected twice with the interval of 21 days between them to 10 participants.
- Adjuvanted PBS: Adjuvanted PBS (Placebo) in the volume of 0.2 ml is injected twice to 10 participants with the interval of 21 days between them.
- Multimeric-001 in PBS 500 mcg: Multimeric-001 in PBS 500 mcg injected twice with the interval of 21 days
- Adjuvanted Multimeric-001 500 mcg: Adjuvanted Multimeric-001 500 mcg injected twice with the interval of 21 days
- Multimeric-001 125 mcg: Multimeric-001 125 mcg in PBS administered once only.
Period: Overall Study
Arm/Group | Multimeric-001 250 mcg in PBS | Adjuvanted Multimeric -001 250 mcg | PBS (Placebo) | Adjuvanted PBS | Multimeric-001 in PBS 500 mcg | Adjuvanted Multimeric-001 500 mcg | Multimeric-001 125 mcg
Started | 10 | 10 | 10 | 10 | 10 | 10 | 3
Completed | 10 | 9 | 10 | 9 | 10 | 9 | 3
Not Completed | 0 | 1 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Multimeric-001 250 mcg in PBS: Multimeric - 001 250 mcg in Phosphate Buffered Solution injected twice with the interval of 21 days between them.
- Total: Total of all reporting groups
Arm/Group | Multimeric-001 250 mcg in PBS | Adjuvanted Multimeric -001 250 mcg | PBS (Placebo) | Adjuvanted PBS | Multimeric-001 in PBS 500 mcg | Adjuvanted Multimeric-001 500 mcg | Multimeric-001 125 mcg | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 3 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 10 | 3 | 63
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (4.0) | 25.8 (8.8) | 25.2 (5.3) | 26.0 (8.4) | 29.0 (7.4) | 25.2 (4.5) | 25.7 (3.3) | 25.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 8 | 9 | 6 | 10 | 3 | 54
  Male | 2 | 0 | 2 | 1 | 4 | 0 | 0 | 9
Region of Enrollment [Number; unit: participants]
  Israel | 10 | 10 | 10 | 10 | 10 | 10 | 3 | 63

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of adverse events per cohort
Time Frame: day 0 until day 42 (termination visit)
Measure: Number; unit: number of reported events
Arm/Group | Multimeric-001 250 mcg in PBS | Adjuvanted Multimeric -001 250 mcg | PBS (Placebo) | Adjuvanted PBS | Multimeric-001 in PBS 500 mcg | Adjuvanted Multimeric-001 500 mcg | Multimeric-001 125 mcg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 3
number of reported events | 46 | 28 | 29 | 36 | 42 | 20 | 2

2. Primary Outcome: Treatment-related Adverse Events
Description: Number of treatment-related adverse events per cohort
Time Frame: Day 0 until day 42 (termination visit)
Measure: Number; unit: number of reported events
Arm/Group | Multimeric-001 250 mcg in PBS | Adjuvanted Multimeric -001 250 mcg | PBS (Placebo) | Adjuvanted PBS | Multimeric-001 in PBS 500 mcg | Adjuvanted Multimeric-001 500 mcg | Multimeric-001 125 mcg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 3
number of reported events | 8 | 11 | 3 | 17 | 3 | 9 | 0

ADVERSE EVENTS:
Time Frame: day 0 until day 42 (termination visit)
Arm/Group | Multimeric-001 250 mcg in PBS | Adjuvanted Multimeric -001 250 mcg | PBS (Placebo) | Adjuvanted PBS | Multimeric-001 in PBS 500 mcg | Adjuvanted Multimeric-001 500 mcg | Multimeric-001 125 mcg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 10/10 | 8/10 | 7/10 | 8/10 | 10/10 | 8/10 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multimeric-001 250 mcg in PBS (N=10) | Adjuvanted Multimeric -001 250 mcg (N=10) | PBS (Placebo) (N=10) | Adjuvanted PBS (N=10) | Multimeric-001 in PBS 500 mcg (N=10) | Adjuvanted Multimeric-001 500 mcg (N=10) | Multimeric-001 125 mcg (N=3)
General disorders (General disorders) | 6 (11) | 3 (7) | 1 (1) | 5 (13) | 4 (9) | 6 (12) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (7) | 3 (10) | 3 (10) | 5 (11) | 2 (6) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations (Investigations) | 4 (6) | 2 (2) | 3 (5) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Metabolism and Nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Musculosceletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 0 (0) | 2 (5) | 2 (2) | 4 (4) | 0 (0)
Nervous system disorders (Nervous system disorders) | 5 (6) | 2 (2) | 2 (3) | 2 (5) | 6 (9) | 3 (4) | 0 (0)
Renal and Urinary disorders (Renal and urinary disorders) | 3 (5) | 2 (4) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (3) | 3 (4) | 4 (8) | 6 (6) | 1 (1) | 0 (0)
Skin and Subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less